CLINICAL TRIAL: NCT06773754
Title: Open-Label Pharmacokinetic Study of Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir Alafenamide Taken as 5 Days Per Week (5/7) Versus Continuous Therapy as 7 Days Per Week (7/7) in HIV-1-Infected Participants Who Are Virally Suppressed
Brief Title: Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir Alafenamide Taken as 5 Days Per Week
Acronym: BICFOTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Visiting staff, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202111050MINB
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Virally Suppressed People With HIV
Keywords: Five-days-On and Two-days-Off; Pharmacokinetic Study; Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir alafenamide; Virally suppressed people with HIV

STUDY DESIGN:
Intervention Model Description: Upon confirmation of eligibility, participants will be randomized in a 1:1 ratio to received 5 days on and 2 days off regimen (5/7 regimen or FOTO group) or continuous therapy (7/7 regimen or Daily group). After 52 weeks, participants in Daily group will be invited to take fixed-dose combination of bictegravir/emtricitabine/tenofovir alafenamide 5 days per week. All participants will be followed for 2 years after enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOTO group (Experimental): Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir alafenamide Taken as 5 Days Per Week (5/7, FOTO group)
  Interventions: Other: Five-days-On and Two-days-Off
- Daily group (No Intervention): Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir alafenamide Taken as 7 Days Per Week (7/7, Daily group)

INTERVENTIONS:
Other: Five-days-On and Two-days-Off — Take Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir alafenamide five days a week (Five-days-On and Two-days-Off)
  Arms: FOTO group

SUMMARY:
The goal of this clinical trial is to learn if fixed-dose combination of bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) taken as 5 days per week (5/7, FOTO group) works well as continuous therapy as 7 days per week (7/7, Daily group) in HIV-1-Infected participants who are virally suppressed. The main questions it aims to answer are:

1. Do the lowest concentrations of BIC at baseline, Week 4, 28, and 52 in the FOTO group achieve the adequate BIC level to control HIV infection?
2. Do the HIV viral loads at Week 4, 28, and 52 remain suppressed in the FOTO group? Researchers will compare FOTO group to Daily group to see if FOTO group can achieve the adequate BIC levels and HIV viral suppression.

Participants will:

1. Take fixed-dose BIC/FTC/TAF 5 days a week or everyday Blood sampling for the lowest concentrations of BIC at baseline, Week 4, 28, and 52
2. Blood sampling for HIV viral loads every 3 months for one year after the enrollment
3. Keep a diary of their drug compliance.
4. Be invited to change to take fixed-dose BIC/FTC/TAF 5 days a week after Week 52 if they are randomised to Daily group initially.
5. Be followed for 2 years after the enrollment.

DETAILED DESCRIPTION:
This protocol describes an open-label, single-center study to evaluate the safety and efficacy of 5/7 intermittent therapy versus 7/7 continuous therapy of coformulated BIC/FTC/TAF FDC in PLWH who are virologically suppressed. The study is comprised of two periods as shown in Figure 1. The first period is an observational 2-week run-in period during which participants who meet the screening criteria will receive daily oral dose of BIC/FTC/TAF. The second study period is a 48-week treatment period (defined as the time the first dose of study drug is administered on Day 1 after randomization through completion of Week 48 assessments) which will evaluate the PK, efficacy, and safety of 5 consecutive days on treatment (typically Monday through Friday) followed by 2 days off treatment (five-on, two-off or 5/7 treatment schedule) regimen compared to continuous therapy (or 7/7) regimen in virologically suppressed HIV-1-infected patients. The study will include Screening of up to 30 days to determine eligibility of participants and to complete disease-related assessments. A self-reported adherence diary will be given to all participants to record whether they take ART during the study period. If the participants in the 5/7 regimen group miss doses during the 5-on days, the missed doses could be taken during the 2-off days to complete the 5 doses a week. Participants will provide written informed consent and visit the study site to complete the screening assessment during the screening period. If the participants are women, contraception is required during study period.

Following successful screening, the 2-week run-in period will commence, during which participants will receive daily coformulated BIC/FTC/TAF dose and only participants with 100% compliance will be eligible to be enrolled in 52-week treatment period. Upon confirmation of eligibility, participants will be randomized in a 1:1 ratio to received 5 days on and 2 days off regimen (5/7 regimen) or continuous therapy (7/7 regimen). Approximately 60 subjects are planned to be randomized. Participants excluded before randomization will be replaced at Screening. After randomization (baseline +/- 1 week), participants will return to the study site at week 4 (+/- 2 weeks) and subsequently every 12 weeks (+/- 3 months) until Week 52 (+/- 1 month) (Table 1). To assess the drug compliance of the study subjects, it is required for them to fill in the paper or online electronic diary cards. Pharmacological study (PK), efficacy and safety assessment will be conducted at Weeks 4, 28 and 52; and QoL will be assessed at baseline and 52 by the electronic form of SF-36v2. The primary endpoint will be assessed at Weeks 4, 28 and 52. Once subjects completed 52-week treatment period, subjects will return to the study site for safety follow-up visit 30 days +/- 3 days after the last dose. If PLWH on 5/7 regimen had virological failure (>1,000 copies/mL) at week 4, 28, or 52, they would be withdrawn from the study. Their HIV isolates would be sent for resistant testing. They would start daily regimen, and their PVL would be checked every 3 months until their PVL return to be suppressed (<200 copies/mL). After Week 52, the participants in continuous therapy (or 7/7) regimen will be invited to change to 5 consecutive days on treatment (typically Monday through Friday) followed by 2 days off treatment (five-on, two-off or 5/7 treatment schedule) regimen. All participants will be followed for 2 years after the enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. PLWH aged 20 years or more
2. PLWH with virological suppression (<50 copies/mL) for 6 months or more
3. PLWH who have received coformulated BIC/FTC/TAF for at least 2 weeks or more

Exclusion Criteria:

1. PLWH with a history of intolerance to antiretroviral regimens containing an integrase inhibitor, ETC/lamivudine, and tenofovir disoproxil fumarate/TAF
2. PLWH with a history of genotypic resistance to integrase inhibitors or TFV
3. PLWH with concurrent use of medications known to pharmacokinetically interact with BIC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BIC trough plasma concentrations | From enrollment to Week 4, 28, and 52 during treatment period
  the proportion of study participants maintaining BIC trough plasma concentrations above the paEC95 of 162 ng/mL after 2 days off coformulated BIC/FTC/TAF at Week 4, 28, and 52 during treatment period

SECONDARY OUTCOMES:
HIV viral suppression | From the enrollment to Week 4, 28, 52, 96 during treatment period
  the proportions of participants with PVL <50 copies/mL at Week 4, 28, and 52 during treatment period and quality of life (QoL) at baseline and Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD would be shared only under requests.

REFERENCES:
- [Derived] Sun HY, Lin YT, Chang WC, Liu WC, Su YC, Kuo CH, Hung CC. Five-days-on-two-days-off (FOTO) versus daily bictegravir/emtricitabine/tenofovir alafenamide in virologically suppressed people with HIV: a pilot randomized clinical trial. J Antimicrob Chemother. 2025 Aug 1;80(8):2179-2186. doi: 10.1093/jac/dkaf186. PMID 40470796